CLINICAL TRIAL: NCT01122862
Title: A Clinical Study to Evaluate the Effect of a Commercial Cosmetic Mouth Rinse on Plaque Re-growth
Brief Title: Effect of a Commercial Cosmetic Mouth Rinse on Plaque Re-growth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Z36420889
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Subjects
Keywords: tooth plaque
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.12% Chlorhexidine Mouthrinse (Active Comparator): Commercially available 0.12% Chlorhexidine mouthrinse
  Interventions: Drug: 0.12% chlorhexidine mouthrinse
- Cosmetic mouthrinse (Active Comparator): Commercially available cosmetic mouthrinse
  Interventions: Other: Cosmetic mouthrinse
- Sterile Water (Placebo Comparator): Sterile Water
  Interventions: Other: Sterile water

INTERVENTIONS:
Drug: 0.12% chlorhexidine mouthrinse — commercially available 0.12% chlorhexidine mouthrinse
  Arms: 0.12% Chlorhexidine Mouthrinse
Other: Cosmetic mouthrinse — Commerically available cosmetic mouthrinse
  Arms: Cosmetic mouthrinse
Other: Sterile water — Sterile water
  Arms: Sterile Water

SUMMARY:
A clinical study to evaluate the effect of a commercial mouth rinse on plaque re-growth

ELIGIBILITY:
Inclusion Criteria:

* Good general and oral health
* At least 20 natural gradable teeth
* Mean plaque score (Turesky Modification of the Quigley Hein Index) of greater than or equal to 2.00 at the first baseline visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Of 31 participants screened, 23 were randomized. 8 enrolled participants were excluded from trial before assignment to groups (3 did not meet the study criterion; remaining 5 were excluded due to other reasons).
Groups:
- Test Mouth Rinse: Participants swirled their oral cavity with 15 milliliters (mL) of commercially available test mouth rinse for 60 seconds and expectorated. Each treatment was administered twice daily for 4 days.
- Chlorhexidine Mouth Rinse (0.12%): Participants swirled their oral cavity with 15 mL of commercially available 0.12% weight by volume (w/v) chlorhexidine mouth rinse for 30 seconds and expectorated. Each treatment was administered twice daily for 4 days.
- Sterile Water: Participants swirled their oral cavity with 15 mL of sterile water for 60 seconds and expectorated. Each treatment was administered twice daily for 4 days.
Period: Period 1
Arm/Group | Test Mouth Rinse | Chlorhexidine Mouth Rinse (0.12%) | Sterile Water
Started | 8 | 8 | 7
Completed | 8 | 7 | 7
Not Completed | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Period: Period 2
Arm/Group | Test Mouth Rinse | Chlorhexidine Mouth Rinse (0.12%) | Sterile Water
Started | 8 (Due to crossover design,a different set of participants received this treatment compared to Period 1) | 7 (Due to crossover design,a different set of participants received this treatment compared to Period 1) | 7 (Due to crossover design,a different set of participants received this treatment compared to Period 1)
Completed | 8 | 7 | 6
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Period: Period 3
Arm/Group | Test Mouth Rinse | Chlorhexidine Mouth Rinse (0.12%) | Sterile Water
Started | 6 (Due to crossover design,a different set of participants received this treatment compared to Period 2) | 7 (Due to crossover design,a different set of participants received this treatment compared to Period 2) | 8 (Due to crossover design,a different set of participants received this treatment compared to Period 2)
Completed | 6 | 7 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants were included for baseline parameters evaluation.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 23
Age Continuous [Mean (Standard Deviation); unit: Years] | 41.9 (14.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 9
Mean Plaque Index Score [Mean (Standard Deviation); unit: Score on a scale] — Plaque scores were assessed using Turesky Modification of the Quigley Hein Index and categorized as 0: No plaque;1: Slight flecks of plaque at the cervical margin of the tooth;2: A thin continuous band of plaque (1 millimeter [mm] or smaller) at the cervical margin of the tooth;3: A band of plaque wider than 1 mm but covering less than 1/3 of the crown of the tooth;4: Plaque covering at least 1/3 but less than 2/3 of the crown of the tooth;5: Plaque covering 2/3 or more of the crown of the tooth. Plaque Index was calculated by taking average of scores over all tooth sites for a participant.
  Score on a scale | 3.01 (0.34)

OUTCOME MEASURES:

1. Primary Outcome: Plaque Index of Test Mouth Rinse Versus Sterile Water After Day 4 of Treatment Administration
Description: Plaque scores were assessed using Turesky Modification of the Quigley Hein Index and categorized as 0: No plaque; 1: Slight flecks of plaque at the cervical margin of the tooth;2: A thin continuous band of plaque (1 mm or smaller) at the cervical margin of the tooth;3: A band of plaque wider than 1 mm but covering less than 1/3 of the crown of the tooth;4: Plaque covering at least 1/3 but less than 2/3 of the crown of the tooth;5: Plaque covering 2/3 or more of the crown of the tooth. The interproximal plaque index was calculated by taking the average of plaque scores over the mesiofacial, distofacial, mesiolingual and distolingual surfaces in the upper and lower jaws for a participant.
Time Frame: Day 4 post treatment administration
Population: Intention to Treat (ITT) population: All randomized participants who received study treatment and had at least one post-baseline efficacy measurement. Due to drop outs, there was difference in number of participants analyzed for this outcome measure. Missing data was not imputed.
Measure: Mean (Standard Error); unit: Score on a scale
Groups:
- Test Mouth Rinse: Participants swirled their oral cavity with 15 mL of commercially available test mouth rinse for 60 seconds and expectorated. Each treatment was administered twice daily for 4 days.
Arm/Group | Test Mouth Rinse | Sterile Water
Number analyzed (Participants) | 22 | 21
Score on a scale | 3.03 (0.10) | 3.23 (0.11)
Statistical Analysis 1: Comparison: Test Mouth Rinse vs Sterile Water; Null hypothesis was no difference between treatments being compared; Test type: Superiority or Other; p = 0.0915, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; ANCOVA with factors for treatment, period and subject (random) with baseline as a covariate; Adjusted Mean Difference = -0.21, 95% CI 2-sided [-0.45 to 0.03] — Difference is first named treatment minus second named treatment such that a negative difference favours the first named treatment

2. Secondary Outcome: Plaque Index Score of Test Mouth Rinse Versus Chlorhexidine Mouth Rinse After Day 4 of Treatment Administration
Description: as for outcome 1
Time Frame: Day 4 post treatment administration
Population: ITT population: All randomized participants who received study treatment and had at least one post-baseline efficacy measurement. Due to drop outs, there was difference in number of participants analyzed for this outcome measure. Missing data was not imputed.
Measure: Mean (Standard Error); unit: Score on a scale
Groups:
- Chlorhexidine Mouth Rinse (0.12% w/v): Participants swirled their oral cavity with 15 mL of commercially available 0.12% w/v chlorhexidine mouth rinse for 30 seconds and expectorated. Each treatment was administered twice daily for 4 days.
Arm/Group | Test Mouth Rinse | Chlorhexidine Mouth Rinse (0.12% w/v)
Number analyzed (Participants) | 22 | 21
Score on a scale | 3.03 (0.10) | 1.36 (0.11)
Statistical Analysis 1: Comparison: Test Mouth Rinse vs Chlorhexidine Mouth Rinse (0.12% w/v); Null hypothesis was no difference in treatments being compared; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; ANCOVA with factors for treatment, period and subject (random) with baseline as a covariate; Adjusted Mean Difference = 1.66, 95% CI 2-sided [1.42 to 1.90] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Plaque Index After 24 Hours of Treatment Administration
Description: as for outcome 1
Time Frame: Day 1 post treatment administration
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Test Mouth Rinse | Chlorhexidine Mouth Rinse (0.12% w/v) | Sterile Water
Number analyzed (Participants) | 22 | 21 | 22
Score on a scale | 1.33 (0.09) | 0.58 (0.09) | 1.29 (0.09)
Statistical Analysis 1: Comparison: Test Mouth Rinse vs Sterile Water; Null hypothesis was no difference between treatments being compared; Test type: Superiority or Other; p = 0.6682, ANCOVA; ANCOVA with factors for treatment, period and subject (random) with baseline as a covariate; Adjusted Mean Difference = 0.04, 95% CI 2-sided [-0.14 to 0.21] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test Mouth Rinse vs Chlorhexidine Mouth Rinse (0.12% w/v); Null hypothesis was no difference between treatments being compared; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment for multiple comparisons was made as the primary comparison was pre-defined; ANCOVA with factors for treatment, period and subject (random) with baseline as a covariate; Adjusted Mean DIfference = 0.74, 95% CI 2-sided [0.57 to 0.92] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Interproximal Plaque Index After Day 4 of Treatment Administration
Description: as for outcome 1
Time Frame: Day 4 post treatment administration
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Test Mouth Rinse | Chlorhexidine Mouth Rinse (0.12% w/v) | Sterile Water
Number analyzed (Participants) | 22 | 21 | 21
Score on a scale | 3.17 (0.10) | 1.48 (0.11) | 3.36 (0.11)
Statistical Analysis 1: Comparison: Test Mouth Rinse vs Sterile Water; Null hypothesis was no difference between treatments being compared; Test type: Superiority or Other; p = 0.1100, ANCOVA — No adjustment for multiple comparisons was made as the primary comparison was pre-defined; ANCOVA with factors for treatment, period and subject (random) with baseline as a covariate; Adjusted Mean Difference = -0.20, 95% CI 2-sided [-0.44 to 0.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test Mouth Rinse vs Chlorhexidine Mouth Rinse (0.12% w/v); Null hypothesis was no difference between treatments being compared; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment for multiple comparisons was made as the primary comparison was pre-defined; ANCOVA with factors for treatment, period and subject (random) with baseline as a covariate; Adjusted Mean Difference = 1.68, 95% CI 2-sided [1.44 to 1.93] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Interproximal Plaque Index After 24 Hours of Treatment Administration
Description: as for outcome 1
Time Frame: Day 1 post treatment administration
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Test Mouth Rinse | Chlorhexidine Mouth Rinse (0.12% w/v) | Sterile Water
Number analyzed (Participants) | 22 | 21 | 22
Score on a scale | 1.60 (0.11) | 0.72 (0.11) | 1.57 (0.11)
Statistical Analysis 1: Comparison: Test Mouth Rinse vs Sterile Water; Null hypothesis was no difference between treatments being compared; Test type: Superiority or Other; p = 0.7280, ANCOVA — No adjustment for multiple comparisons was made as the primary comparison was pre-defined; ANCOVA with factors for treatment, period and subject (random) with baseline as a covariate; Adjusted Mean Difference = 0.03, 95% CI [-0.16 to 0.23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test Mouth Rinse vs Chlorhexidine Mouth Rinse (0.12% w/v); Null hypothesis was no difference between treatments being compared; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment for multiple comparisons was made as the primary comparison was pre-defined; ANCOVA with factors for treatment, period and subject (random) with baseline as a covariate; Adjusted Mean Difference = 0.88, 95% CI 2-sided [0.68 to 1.08] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: All adverse events encountered or spontaneously reported following administration of any investigational product (including washout product), or for up to 5 days after the last administration of investigational product were recorded.
Arm/Group | Test Mouth Rinse | Chlorhexidine Mouth Rinse (0.12% w/v) | Sterile Water
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 1/22 | 1/22 | 2/22
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Mouth Rinse (N=22) | Chlorhexidine Mouth Rinse (0.12% w/v) (N=22) | Sterile Water (N=22)
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Multiple Sclerosis Relapse (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.